CLINICAL TRIAL: NCT02490488
Title: Phase 2/3 Study of Masitinib in Combination With Gemcitabine Versus Gemcitabine Alone in Advanced/Metastatic Epithelial Ovarian Cancer Patients in Second Line Being Refractory to First Line Platinum Treatment or in Third Line
Brief Title: Masitinib in Combination With Gemcitabine in Advanced/Metastatic Epithelial Ovarian Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB12008
Record Dates: First submitted 2015-05-18; First posted 2015-07-03 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; tyrosine kinase inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — masitinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Masitinib & gemcitabine (Experimental): Participants receive masitinib (6 mg/kg/day), given orally twice daily, plus gemcitabine 1000 mg/m² administered by 30 minutes infusion once a week during 3 weeks followed by 1 week without infusion.
  Interventions: Drug: Masitinib; Drug: Gemcitabine
- Placebo & gemcitabine (Placebo Comparator): Participants receive placebo (6 mg/kg/day), given orally twice daily, plus gemcitabine 1000 mg/m² administered by 30 minutes infusion once a week during 3 weeks followed by 1 week without infusion.
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Masitinib & gemcitabine
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo & gemcitabine

SUMMARY:
The objective is to evaluate the efficacy and safety of masitinib in combination with gemcitabine in refractory ovarian cancer patients.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor that is thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment. The objective of this study is to evaluate the efficacy and safety of masitinib in combination with gemcitabine as compared with single agent gemcitabine in advanced or metastatic epithelial ovarian cancer patients who are refractory to platinum treatment. This is an open-label, randomized, active-controlled, phase 2/3 study. The study's primary efficacy measure will be overall survival. Masitinib will be prescribed until disease progression (or treatment switch to next line of treatment), death, limiting toxicity or patient consent withdrawal. The study design is a two-stage adaptive design, meaning that it includes a prospectively planned opportunity for modification of one or more specified aspects of the study (for example patient enrollment).

ELIGIBILITY:
Main inclusion criteria:

1. Female patient, with histologically or cytologically confirmed advanced / metastatic epithelial ovarian cancer (including primary peritoneal and primary fallopian tube cancer), which is either:

   * First line platinum-refractory ovarian cancer (progression during first-line platinum-based chemotherapy)
   * First line platinum-resistant ovarian cancer (relapsing within 6 months after the end of first-line chemotherapy);
   * Candidate to third line of treatment (refractory, resistant, or sensitive to 2nd line platinum-based therapy or patients who progressed after other type of chemotherapy in 2nd line).
2. Patient with adequate organ function per laboratory tests evaluations

Main exclusion criteria:

1. Patient intolerant to gemcitabine
2. Patient who has not recovered from any significant treatment toxicities prior to baseline (≥Grade 2)
3. Pregnant or nursing female patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

SECONDARY OUTCOMES:
Overall Progression Free Survival (PFS) | From day of randomization to disease progression or death, assessed for a maximum of 60 months
  Progression Free Survival (PFS) [Time Frame: From day of randomization to disease progression or death, assessed for a maximum of 60 months] Progression Free Survival is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed by CT scan according to RECIST criteria recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Grenier, Dr, Principal Investigator — AB Science
Locations (6):
- Centre hospitalo-universitaire de Beni Messous, Algiers, Algeria
- Institut Sainte Catherine, Avignon, France
- City Oncology Clinic, Saint Petersburg, Russia
- Complejo Hospitalario Universitario de Santiago, Santiago, Spain
- Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv, Ukraine
- University Hospital Coventry, Coventry, United Kingdom